CLINICAL TRIAL: NCT06285539
Title: Drug Rediscovery for Rare Immune Mediated Inflammatory Diseases
Acronym: DRIMID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Alfasigma S.p.A. (Industry); ReumaNederland (Unknown); Autoimmune Research and Collaboration Hub (Unknown)
Responsible Party: Principal Investigator, Jacob M van Laar, Prof. dr., UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-502968-20
Record Dates: First submitted 2024-02-12; First posted 2024-02-29 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Behcet's Disease; Idiopathic Inflammatory Myopathies; IgG4-related Disease
Keywords: JAK-inhibition
MeSH Terms: conditions — Behcet Syndrome; Myositis; Immunoglobulin G4-Related Disease | interventions — GLPG0634

STUDY DESIGN:
Intervention Model Description: A 26-week multicenter, open-label, uncontrolled, non-randomized, non-blinded proof-of-concept, two-stage phase 2 study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): 26 weeks of Filgotinib once daily, 200mg, orally,
  Interventions: Drug: Filgotinib

INTERVENTIONS:
Drug: Filgotinib — Filgotinib

SUMMARY:
Research into novel therapies for rare, immune-mediated inflammatory diseases (IMIDs) is limited due to small patient populations. Patients with Behçet's disease (BD), idiopathic inflammatory myopathy (IIM, also known as myositis) and IgG4-related disease (IgG4-RD) are treated with high-dosed glucocorticoids, methotrexate, azathioprine and mycophenolate mofetil, mostly for long periods of time with attendant risks of long-term toxicity, including infections. Therefore, there is an urgent need for new, more specific anti-inflammatory therapies such as targeted synthetic and biological disease-modifying antirheumatic drugs. Due to the role of type 1 interferon in both BD, IIM and IgG4-RD, JAK-STAT inhibition may be a promising treatment strategy in these conditions, because JAK1 is critical for the signal transduction of pro-inflammatory cytokine receptors. Previous research showed that JAK1 inhibition reduces activation of type 1 interferon-regulated proteins and key chemokines that control tissue inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of older
* One of the following rare IMIDs:

  * Diagnosis of Behçet's disease without refractory life, organ or sight-threatening symptoms with active disease, defined as a BDCAF >2 (new BDCAF) or >15 (old BDCAF) or with active disease, based on clinical grounds (e.g. the need to start new or additional medication
  * Diagnosis of idiopathic inflammatory myopathy, according to diagnostic criteria:

Dermatomyositis: Dermatomyositis Classification Criteria according to the European Neuromuscular Centre guidelines 201852 or anti-synthetase syndrome: Anti- synthetase syndrome Classification Criteria according to the European Neuromuscular Centre guidelines 200353, both with active disease, defined as a CDASI score of ≥5 or abnormal levels of at least 1 of the following enzymes: creatine kinase (≥ 4× upper limit of normal [ULN]), aldolase (≥4 × ULN), lactate dehydrogenase (LDH ≥4 × ULN), aspartate transaminase (AST ≥4 × ULN), alanine aminotransferase (ALT ≥4 × ULN) or a MRI within the last 3 months indicative of active inflammation (e.g. edema signal pattern in affected proximal muscles) or active disease based on clinical grounds, e.g. the need to start new or additional medication

* Diagnosis of IgG4-related disease, according to 2019 ACR/EULAR guidelines, with active disease, defined as: IgG4-related disease responder index >10 or active disease based on clinical grounds, e.g. the need to start new or additional medication

  * Refractory disease, defined as symptomatic disease that persists despite a 12-week trial of glucocorticoid therapy as well as lack of response to at least one other immunosuppressive agent such as methotrexate (MTX), mycophenolate mofetil (MMF), azathioprine (AZA) or rituximab or intolerance to standard-of-care treatment, as defined by the treating physician.
  * No evidence of active or latent or inadequately treated infection with mycobacterium tuberculosis (TB) as defined by all of the following: both a negative QuantiFERON-TB Gold (QFT-G) In-Tube test and a Mantoux tuberculin skin test performed at or within 3 months prior to screening and no signs suggestive of active TB infection as determined (and documented) by a qualified radiologist or pulmonologist as per local standard of care on a chest radiograph and no history of either untreated or inadequately treated latent or active TB infection.

Exclusion Criteria:

* Age <18 years
* Age ≥65 years
* Life expectancy less than 6 months
* Juvenile DM, myositis overlapping with other autoimmune diseases, immune mediated necrotizing myopathy (IMNM), inclusion-body myositis or cancer-associated myositis
* End-stage IIM wherein muscle weakness is most likely due to muscle damage, rather than myositis disease activity
* Increased risk of major cardiovascular problems
* Current smoker or smoked for a long time in the past
* Pregnancy or lactation
* Previous use of other JAK inhibitors
* Use of any investigational drug within one month prior to screening or within five half-lives of the investigational agent, whichever is longer.
* Human Immunodeficiency Virus (HIV) infection
* Presence of an active infection or viral hepatitis type B or C
* History of shingles or recurrent herpes simplex infection
* Concomitant malignancies or previous malignancies within the last five years (with exception of adequately treated basal or squamous cell carcinoma of the skin)
* Increased risk of cancer
* Kidney injury with estimated glomerular filtration rate <15mL/min/1.73m2
* Liver failure Child Pugh C
* Absolute neutrophil count <1*109
* Absolute leukocyte count <0.5*109
* Hemoglobin <5mmol/L - Inability to comply with study and/or follow-up procedures
* Known recent substance abuse (drugs or alcohol).
* Poor tolerability of venipuncture or lack of adequate venous access for required blood sampling during the study period.
* Previous non-adherence to immunosuppressants
* Hypersensitivity to the active substance or to any of the excipients
* Rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
EQ-5D-5L | 26 weeks
  Change from baseline in EuroQoL-5D-5L
Disease activity in Behcet's patients | 26 weeks
  Change from baseline in Behcet's Disease Current Activity Form (BDCAF)
Disease activity in myositis patients | 26 weeks
  Change from baseline in Total Improvement Score (TIS) of the International Myositis Assessment Clinical Studies (IMACS) group
Disease activity in IgG4-RD patients | 26 weeks
  Change from baseline in IgG4-RD responder index

SECONDARY OUTCOMES:
Corticosteroid toxicity | 26 weeks
  Change from baseline in Glucocorticoid Toxicity Index (GTI)
Corticosteroid dosage | 26 weeks
  Change from baseline in glucocorticoid dose
VAS score of pain | 26 weeks
  Change from baseline in pain scores on the Visual Analog Scale (0-100mm). A higher score is a worse outcome
Fatigue | 26 weeks
  Change from baseline in fatigue scores on the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F). A higher score is a worse outcome
Treatment-related adverse events | 26 weeks
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Jaap M van Laar, Prof. dr., Principal Investigator — UMC Utrecht
Locations (6):
- Netherlands (6):
  - Amsterdam UMC, Amsterdam
  - Zuyderland Medical Center, Heerlen
  - Radboud university medical center, Nijmegen
  - Erasmus MC, Rotterdam
  - Hagaziekenhuis, The Hague
  - University Medical Center, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Geertsema-Hoeve BC, van Laar JAM, Raaphorst J, Tas SW, Welsing PMJ, Goekoop RJ, Checa CM, Thurlings RM, Rekers NH, Present E, van Laar JM. Multicentre, 26-week, open-label phase 2 trial of the JAK inhibitor filgotinib in Behcet's disease, idiopathic inflammatory myopathies and IgG4-related disease: DRIMID study protocol. BMJ Open. 2025 Feb 6;15(2):e089827. doi: 10.1136/bmjopen-2024-089827. PMID 39915014